CLINICAL TRIAL: NCT04210466
Title: COMP.ACT: Testing the Effect of Explicit Self-compassion Exercises in an ACT Group Intervention for Chronic Pain
Brief Title: COMP.ACT for Chronic Pain Exercises in an ACT Group Intervention for Chronic Pain
Acronym: COMPACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Sérgio Andrade Carvalho, Principal Investigator, University of Coimbra
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFRH/BD/112833/2015
Record Dates: First submitted 2019-12-18; First posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Chronic Pain
Keywords: chronic pain; Acceptance and Commitment Therapy (ACT); Compassion
MeSH Terms: conditions — Chronic Pain | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance & Commitment Therapy + Compassion (COMP.ACT) (Experimental): an ACT intervention + 2 sessions of explicit self-compassion meditation exercises.
  Interventions: Behavioral: Acceptance & Commitment Therapy + Compassion (COMP.ACT)
- Acceptance & Commitment Therapy (ACT) (Active Comparator): an ACT intervention + 2 Q&A sessions.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)

INTERVENTIONS:
Behavioral: Acceptance & Commitment Therapy + Compassion (COMP.ACT) — 8 sessions, 2h each. Intervention includes meditation exercises, behavioral exercises, group discussions, and the structure is the following Session 1: INTRODUCTION: control is the problem Session 2: THE BODY AS PRESENT: promoting body awareness through mindfulness Session 3: COMPASSION I: from self-criticism to self-care Session 4: COMPASSION II: the body as an anchor to self-compassion Session 5: ACCEPTANCE: there is more to accept than just pain Session 6: (RE)DISCOVERING VALUES: in search of a valued life Session 7: ACT NOW: from values to committed action Session 8: CARRY ON AFTER COMP.ACT: program summary
  Arms: Acceptance & Commitment Therapy + Compassion (COMP.ACT)
Behavioral: Acceptance and Commitment Therapy (ACT) — 8 sessions, 2h each. Intervention includes meditation exercises, behavioral exercises, group discussions, and the structure is the following Session 1: INTRODUCTION: control is the problem Session 2: THE BODY AS PRESENT: promoting body awareness through mindfulness Session 3: Q&A 1 Session 4: Q&A 2 Session 5: ACCEPTANCE: there is more to accept than just pain Session 6: (RE)DISCOVERING VALUES: in search of a valued life Session 7: ACT NOW: from values to committed action Session 8: CARRY ON AFTER COMP.ACT: program summary
  Arms: Acceptance & Commitment Therapy (ACT)

SUMMARY:
This study tests the efficacy of adding explicit self-compassion meditation exercises in an ACT intervention for chronic pain (COMP.ACT). COMP.ACT is an 8-session, 2h each, psychological intervention for women with chronic pain. Half of participants will receive an ACT intervention + 2 Q&A sessions, and half of participants will receive an ACT intervention + 2 compassion-focused sessions with explicit self-compassion exercises.

DETAILED DESCRIPTION:
Acceptance and Commitment Therapy (ACT) is a transdiagnostic approach, with empirical support in adapting to several chronic health conditions, such as chronic pain (CP), and its main purpose is to improve functioning and decrease interference of pain with valued life goals. Although the American Psychological Association (APA) has stated ACT as having empirical support in CP (http://www.div12.org/PsychologicalTreatments/treatments/chronicpain_act.html), with several studies showing its efficacy, there is still room for improvement. This might be attained by adding theoretically compatible components such as self-compassion. Although ACT has recently incorporated self-compassion as one of its outcomes, this has not been considered in any ACT intervention study for CP. Compassion-based approaches has been effective in targeting self-criticism, and has been effective in reducing a large array of psychopathological symptoms that are also common in CP (e.g. depression and anxiety). The current study aims to test the adding value of explicit self-compassion exercises in an ACT group intervention for CP.

General study design Participants previously diagnosed with CP by a physician will be assigned into two different conditions/groups: a group intervention for CP that includes explicit self-compassion exercises (COMP.ACT); and a group intervention that does not include explicit self-compassion exercises (ACT). The efficacy of COMP.ACT will be assessed by comparing it with the ACT condition.

Sample This study aims to focus on musculoskeletal CP as it is the most common cause of CP. Also, the study will recruit women with CP. Patients will be provided a study description, a consent form and the research team contact for further clarifications.

The COMP.ACT protocol has the following goals: (a) promote engagement in meaningful and effective activities, even with pain and distress, (b) improving present-focused awareness and acceptance of thoughts, feelings, and physiological sensations; (c) developing a self-compassion stance towards personal difficulties, and (d) promote commitment and engagement with valued actions.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain diagnosis(es),
* age between 18-65,
* residence in center region of Portugal,
* Availability to attend sessions.

Exclusion Criteria:

* Symptoms of psychosis,
* Non-suicidal self-injury,
* Suicide ideation,
* Severe Depression,
* Substance Abuse.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
change from Numeric Pain Rating Scale at 2 months (post-intervention) | baseline, at 2 months (post-intervention)
  Pain intensity - higher scores mean more pain intensity
change from Pain Disability Index | baseline, 2 months (post-intervention), 6 months (follow-up)
  Pain disability - higher scores mean more pain disability
change from World Health Organization Quality of Life - Bref | baseline, 2 months (post-intervention), 6 months (follow-up)
  Quality of Life - higher scores mean more quality of life
change from Depression Anxiety and Stress Scale - 21 items | baseline, 2 months (post-intervention), 6 months (follow-up)
  Depression, anxiety and stress symptoms - higher scores mean more depression, anxiety and stress symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio Carvalho, Principal Investigator — CINEICC - University of Coimbra
Locations (1):
- Consulta da dor, Serviço de Anestesiologia, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No